CLINICAL TRIAL: NCT00387660
Title: Phase II Study of Irinotecan and Carboplatin in Metastatic or Relapsed Small-Cell Lung Cancer
Brief Title: Irinotecan and Carboplatin in Treating Patients With Metastatic or Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC-124; 200210637 (Other: UC Davis); PFIZER-Z1000752 (Other Grant/Funding Number: Pfizer); P30CA093373 (NIH); NCT00462800 (obsolete NCT alias)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Carboplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metastatic SCLC (Experimental): Irinotecan 200 mg/m2, every 21 days (intravenous) + Carboplatin AUC = 5 mg/ml x min (intravenous), every 21 days for 6 cycles
  Interventions: Drug: carboplatin; Drug: irinotecan
- Relapsed SCLC (Experimental): Irinotecan 150 mg/m2 (intravenous), every 21 days + Carboplatin AUC = 5 mg/ml x min (intravenous, every 21 days for 6 cycles
  Interventions: Drug: carboplatin; Drug: irinotecan

INTERVENTIONS:
Drug: carboplatin — Patients receive carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Paraplatin; Paraplatin-AQ
Drug: irinotecan — Patients receive irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Camptosar®; Camptothecin-11; CPT-11

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with carboplatin works in treating patients with metastatic or recurrent small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rates in patients with metastatic or recurrent small cell lung cancer treated with irinotecan hydrochloride and carboplatin.
* Determine the median survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (yes vs no) and disease stage (metastatic vs relapsed).

Patients receive irinotecan hydrochloride IV over 90 minutes and carboplatin IV over 15-30 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer, meeting 1 of the following criteria:

  * Previously untreated metastatic or extensive disease

    * Malignant pleural effusion or multifocal lung disease is considered metastatic or extensive disease
    * Prior radiotherapy allowed
  * Recurrent disease

    * Limited, metastatic, or extensive disease
    * Relapsed after prior chemotherapy, excluding irinotecan hydrochloride

      * At least 90 days since prior chemotherapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 1 cm by physical examination or radiographic techniques
* Known brain metastases allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* White Blood Cells > 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ 1.5 mg/dL
* SGOT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No medical disease that, in the opinion of the investigator, would preclude study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 10 days since prior radiotherapy (including brain)
* No prior irinotecan hydrochloride
* At least 2 weeks since prior and no concurrent anticonvulsants
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-10; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derick H. Lau, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Result] Chen G, Huynh M, Fehrenbacher L, West H, Lara PN Jr, Yavorkovsky LL, Russin M, Goldstein D, Gandara D, Lau D. Phase II trial of irinotecan and carboplatin for extensive or relapsed small-cell lung cancer. J Clin Oncol. 2009 Mar 20;27(9):1401-4. doi: 10.1200/JCO.2008.20.2127. Epub 2009 Feb 9. PMID 19204194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was 6 years. Subjects were recruited at 4 large medical centers.
Groups:
- Arm A - Metastatic SCLC (no Previous Chemo): Extensive small cell lung cancer with no previous chemotherapy
- Arm B - Relapsed SCLC (Previous Chemo): Relapsed small cell lung cancer with previous chemotherapy
Period: Overall Study
Arm/Group | Arm A - Metastatic SCLC (no Previous Chemo) | Arm B - Relapsed SCLC (Previous Chemo)
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Metastatic small cell lung cancer with no previous chemotherapy
- Arm B: Relapsed small cell lung cancer with previous chemotherapy
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: years] | 67 [50 to 81] | 65 [43 to 80] | 65 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 22 | 17 | 39
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria for target lesions and assessed by radiographic techniques. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Population: All participants for whom response evaluation measurements were recorded at Baseline and after 2 cycles.
Measure: Number; unit: percentage of participants
Groups:
- Arm A: Irinotecan (200 mg/m2, q21 days) for 6 cycles, Carboplatin (AUC=5mg/ml x min, q21 days) for 6 cycles
- Arm B: Irinotecan (150 mg/m2, q21 days) for 6 cycles, Carboplatin (AUC=5mg/ml x min, q21 days) for 6 cycles
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 34 | 38
percentage of participants | 65 | 50

2. Secondary Outcome: Median Survival of Patients Treated With This Regimen
Description: The length of time from the start of treatment that half of the patients in a group of patients diagnosed with the disease are still alive.
Time Frame: Up to 36 months
Population: All participants for whom response evaluation measurements were recorded at Baseline and after 2 cycles.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 34 | 38
months | 10 [6 to 14] | 10 [6 to 14]

3. Secondary Outcome: Number of Participants With Toxicity
Description: All adverse events were graded according to the National Cancer InstituteCommon Toxicity Criteria, version 2.0. All 80 patients were assessable for toxicity at least for the first cycle.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 40 | 40
Participants | 40 | 40

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 2/40 | 2/40
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=40) | Arm B (N=40)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=40) | Arm B (N=40)
Neutropenia (Blood and lymphatic system disorders) | 21 | 22
Neutropenic fever (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 9
Anemia (Blood and lymphatic system disorders) | 4 | 6
Diarrhea (Gastrointestinal disorders) | 9 | 8
Nausea/emesis (Gastrointestinal disorders) | 3 | 5
Treatment-related death (Infections and infestations) | 2 | 1 — Succumbed to sepsis in the setting of neutropenia

LIMITATIONS AND CAVEATS:
Of the 80 patients, 72 were assessable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes